CLINICAL TRIAL: NCT05170477
Title: Influence of Apical Patency Concept Upon Postoperative Pain After Root Canal Treatment in Molars With Pulpal Disease. A Randomized Controlled Clinical Trial.
Brief Title: Influence of Apical Patency Concept Upon Postoperative Pain After Root Canal Treatment
Acronym: patency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Heba Elasfouri, Associate professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Endo 27-11-2021
Record Dates: First submitted 2021-11-27; First posted 2021-12-28 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Apical aptency (Experimental): In Gp A, apical patency will be maintained till obturation using electronic apex locator confirmed radiographically
  Interventions: Procedure: apical patency
- Non-apical patency (Active Comparator): in Gp B apical patency will not be maintained
  Interventions: Procedure: Non-apical surgery

INTERVENTIONS:
Procedure: apical patency — In Gp A, apical patency will be maintained till obturation using electronic apex locator confirmed radiographically. Finally, Root canals will be obturated using cold lateral compaction technique. The molars will be permanently restored using composite resin restoration and will be scheduled for extra coronal restoration.
  Arms: Apical aptency
Procedure: Non-apical surgery — in Gp B apical patency will not be maintained. Finally, Root canals will be obturated using cold lateral compaction technique. The molars will be permanently restored using composite resin restoration and will be scheduled for extra coronal restoration
  Arms: Non-apical patency

SUMMARY:
The aim of this clinical study is to evaluate the influence of apical patency concept implementation upon postoperative pain following root canal treatment in a single visit approach in molars with pulpal disease.

DETAILED DESCRIPTION:
All patients will be treated in a single session approach regardless of the group. All molars will be anesthetized either through infiltration in case of maxillary molars or inferior alveolar nerve block in case of mandibular molars using Octocaine 2% with epinephrine 1: 100,000 (Lidocaine HCl, Novocol Pharmaceutical, Ontario, Canada.). Rubber dam will be applied; and access will be opened using Endo access bur.

Canals will be scouted using manual patency file in a watch winding maneuver and then coronal flaring will be performed using Gates Glidden drill #3 in a brushing motion away from dangerous zone. Root canals will be copiously irrigated using 10 ml 2.5% sodium hypochlorite NaOCl (Clorox; Egyptian Company for household bleach, Egypt) delivered using 28 Gauge safety Steri Irrigation Tip (DiaDent Group International, Burnaby, BC, Canada) inserted 3 mm below cementoenamel junction. Working length will be determined using electronic apex locator Root ZX II (J. Morita Mfg. Corp, Kyoto, Japan) and confirmed radiographically using parallel technique with receptor holding device. Canals will be irrigated again with 10ml 1.5% NaOCl, which will be delivered 2mm coronal to apical canal terminus. Irrigation will be hydro-dynamically agitated with EndoActivator device (Dentsply Maillefer, Baillagues, Switzerland) using yellow tips #20/06 inserted 2mm short of working length for 60 seconds. Root canals will be shaped using ProTaper next rotary Ni-Ti files (Dentsply Maillefer, Baillagues, Switzerland). In Gp A, apical patency will be maintained till obturation using electronic apex locator confirmed radiographically while in Gp B apical patency will not be maintained. Finally, Root canals will be obturated using cold lateral compaction technique. The molars will be permanently restored using composite resin restoration and will be scheduled for extra coronal restoration.

ELIGIBILITY:
Inclusion Criteria:

* •1. Patient age between 18-60 years old.

  * 2. Both males and females will be included.
  * 3. All patients are in a good health without systemic condition.
  * 4. The offending tooth is a molar.
  * 5. The offending molar is indicated for root canal treatment.
  * 6. One molar for every patient.
  * 7. All patients will sign an informed consent.

Exclusion Criteria:

* 1. The offending tooth has previous attempt of pulp therapy or root canal treatment.

  * 2. The patient showing any clinical or radiographic evidence of periapical pathosis.
  * 3. Patients received analgesics or systemic antibiotic prior to treatment.
  * 4. Immunocompromised patients.
  * 5. Any unknown infectious disease (e.g. HBV, HCV, HIV, or T.B.)
  * 6. History of cancer with radio or chemotherapy.
  * 7. Offending molar with mobility score ≥2.
  * 8. Offending molar with pocket depth ≥6mm.
  * 9. Immature molars.
  * 10. Nonodontogenic pain.
  * 11. Patients with more than one tooth requiring endodontic intervention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
postoperative pain intensity using numerical rating scale | after 6 hours after root canal treatment
  postoperative pain after root canal treatment
postoperative pain intensity using numerical rating scale | after12 hours after root canal treatment
  postoperative pain after root canal treatment
postoperative pain intensity using numerical rating scale | after 24 hours after root canal treatment
  postoperative pain after root canal treatment
postoperative pain intensity using numerical rating scale | after 48 hours after root canal treatment
  postoperative pain after root canal treatment

CONTACTS AND LOCATIONS:
Overall Officials: Heba A ElAsfouri, AssProfessor, Study Director — Cairo University
Locations (1):
- Heba ahmed ElAsfouri, Giza, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] al-Omari MA, Dummer PM. Canal blockage and debris extrusion with eight preparation techniques. J Endod. 1995 Mar;21(3):154-8. doi: 10.1016/s0099-2399(06)80443-7. PMID 7561660